CLINICAL TRIAL: NCT02403830
Title: Effect of the Peripheral Opioid Receptor Antagonist Methylnaltrexone on the Pharmacokinetic and Pharmacodynamic Profiles of Ticagrelor in Patients Receiving Morphine: a Prospective, Randomized Placebo-controlled Trial
Brief Title: Effect of Methylnaltrexone on the PK/PD Profiles of Ticagrelor in Patients Treated With Morphine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AZ 10583 IISR
Record Dates: First submitted 2015-02-17; First posted 2015-03-31 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — methylnaltrexone; Morphine; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylnaltrexone (Experimental): Patients will be randomly assigned in a 1:1 fashion to receive either i.v methylnaltrexone or placebo (0.9% sodium chloride iv injection). Methylnaltrexone, at a dose of 0.3 mg/Kg, will be administered diluted with 5 ml of normal saline as a single i.v. bolus over 1 minute followed by morphine (5-mg intravenous bolus). Then patients will receive iv morphine and a loading dose of ticagrelor.
  Interventions: Drug: Methylnaltrexone; Drug: Morphine; Drug: Ticagrelor
- Placebo (Placebo Comparator): Patients will be randomly assigned in a 1:1 fashion to receive either i.v methylnaltrexone or placebo (0.9% sodium chloride iv injection). Methylnaltrexone, at a dose of 0.3 mg/Kg, will be administered diluted with 5 ml of normal saline as a single i.v. bolus over 1 minute followed by morphine (5-mg intravenous bolus). Then patients will receive iv morphine and a loading dose of ticagrelor.
  Interventions: Other: Placebo; Drug: Morphine; Drug: Ticagrelor

INTERVENTIONS:
Drug: Methylnaltrexone — Methylnaltrexone will be administered diluted with 5 ml of normal saline as a single iv bolus
  Other Names: Relistor
  Arms: Methylnaltrexone
Other: Placebo — Placebo will be administered as a 0.9% sodium chloride iv injection
  Arms: Placebo
Drug: Morphine — After methylnaltrexone, patients will receive 5-mg intravenous morphine
  Other Names: Morphine sulfate
Drug: Ticagrelor — After morphine administration, patients will receive a 180-mg ticagrelor loading dose
  Other Names: Brilinta

SUMMARY:
Ticagrelor is associated with more prompt and potent antiplatelet effects compared with clopidogrel, leading to better clinical outcomes, including reduced cardiovascular mortality, across the spectrum of patients with acute coronary syndrome, including those with ST-elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI). However, in this latter setting a delay in the onset of its antiplatelet effects has been shown. Morphine has been identified as a cause of delayed P2Y12 inhibition in patients with STEMI. Methylnaltrexone is a parenteral peripheral opioid receptor antagonist which has the potential to prevent or reverse opioid-induced peripherally mediated side effects without affecting analgesia. However, whether the use of intravenous methylnaltrexone may overcome the effects of morphine administration on the pharmacokinetic (PK) and pharmacodynamics (PD) profiles of ticagrelor has not been investigated yet. The proposed investigation will include patients with coronary artery disease and will have a prospective, randomized, cross-over design.

DETAILED DESCRIPTION:
Ticagrelor is associated with more prompt and potent antiplatelet effects compared with clopidogrel, leading to better clinical outcomes, including reduced cardiovascular mortality, across the spectrum of patients with acute coronary syndrome, including those with ST-elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI). However, in this latter setting a delay in the onset of its antiplatelet effects has been shown. Morphine has been identified as a cause of delayed P2Y12 inhibition in patients with STEMI. In fact, opiates are known to inhibit gastric emptying, leading to delayed absorption and potentially decreasing peak plasma levels of orally administered drugs. Methylnaltrexone is a parenteral peripheral opioid receptor antagonist which has the potential to prevent or reverse opioid-induced peripherally mediated side effects (i.e. gastric emptying inhibition) without affecting analgesia. Studies have shown that methylnaltrexone effectively prevented morphine-induced gut motility change. However, whether the use of intravenous methylnaltrexone may overcome the effects of morphine administration on the pharmacokinetic (PK) and pharmacodynamics (PD) profiles of ticagrelor has not been investigated yet. The proposed investigation will include patients with coronary artery disease and will have a prospective, randomized, cross-over design. Patients will be randomized to receive either intravenous methylnaltrexone or placebo. Immediately after methylnaltrexone administration, patients will receive intravenous morphine and then will receive a 180-mg ticagrelor loading dose 15 minutes after morphine administration. After a 7 ± 2 days wash-out period, patients will cross-over to the alternate study-treatment arm. At each visit, blood samples for PK and PD assessments will be collected at several time points. This study will provide insights on a possible treatment strategy to overcome the impaired P2Y12 inhibition induced by morphine.

ELIGIBILITY:
Inclusion criteria:

* Patients with angiographically documented CAD.
* On treatment with low-dose aspirin (81 mg) for at least 30 days, as per standard of care.
* Age between 18 and 80 years old.

Exclusion criteria:

* History of prior intracranial bleeding.
* On treatment with a P2Y12 receptor antagonist (ticlopidine, clopidogrel, prasugrel, ticagrelor) or with vorapaxar in past 30 days.
* Known allergies to ticagrelor.
* On treatment with any oral anticoagulant (vitamin K antagonists, dabigatran, rivaroxaban, apixaban).
* Treatment with glycoprotein IIb/IIIa inhibitors in past 7 days.
* Known blood dyscrasia or bleeding diathesis.
* Platelet count <80x106/mL.
* Hemoglobin <10 g/dL.
* Active bleeding.
* Hemodynamic instability.
* Creatinine clearance <30 mL/minute (as estimated by Cockcroft-Gault formula).
* Severe hepatic dysfunction.
* Acute or severe bronchial asthma or upper airway obstruction.
* Known or suspected mechanical gastrointestinal obstruction.
* Patients with sick sinus syndrome (SSS) or high degree AV block without pacemaker protection.
* Current treatment with any drug interfering with morphine: central nervous system depressants (other narcotic analgesics, general anesthetics, phenothiazines, tricyclic antidepressants, tranquilizers, sedatives, hypnotics, antiemetics, and alcohol), muscle relaxants, mixed agonist/antagonist analgesics (i.e., pentazocine, nalbuphine, and butorphanol), cimetidine, monoamine oxidase inhibitors (MAOIs), anticholinergics.
* Current treatment with drugs interfering with CYP3A4 metabolism (to avoid interaction with ticagrelor): Ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and telithromizycin.
* Pregnant females*. *Women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Angiolillo, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franchi F, Rollini F, Park Y, Hu J, Kureti M, Rivas Rios J, Faz G, Yaranov D, Been L, Pineda AM, Suryadevara S, Soffer D, Zenni MM, Bass TA, Angiolillo DJ. Effects of Methylnaltrexone on Ticagrelor-Induced Antiplatelet Effects in Coronary Artery Disease Patients Treated With Morphine. JACC Cardiovasc Interv. 2019 Aug 26;12(16):1538-1549. doi: 10.1016/j.jcin.2019.05.028. Epub 2019 Jul 31. PMID 31377269

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2015 and April 2016 a total of 34 patients were recruited and consented at the University of Florida Health Science Center at UF Health Jacksonville - Division of Cardiology.
Pre-assignment Details: Four subjects withdrew their consent before randomization and did not receive study drug. Therefore a total of 30 patients were randomized.
Groups:
- Methylnaltrexone First: Patients were randomly assigned in a 1:1 fashion to receive either i.v methylnaltrexone or placebo (0.9% sodium chloride iv injection). Methylnaltrexone, at a dose of 0.3 mg/Kg, was administered diluted with 5 ml of normal saline as a single i.v. bolus over 1 minute followed by morphine (5-mg intravenous bolus). Then patients received iv morphine and a loading dose of ticagrelor. In this arm patients received methylnaltrexone at visit 1. After a 7 ± 2 days wash-out period, patients crossed-over to the alternate study-treatment arm (placebo).
  Methylnaltrexone: Methylnaltrexone will be administered diluted with 5 ml of normal saline as a single iv bolus
  Morphine: After methylnaltrexone, patients will receive 5-mg intravenous morphine
  Ticagrelor: After morphine administration, patients will receive a 180-mg ticagrelor loading dose
- Placebo First: Patients were randomly assigned in a 1:1 fashion to receive either i.v methylnaltrexone or placebo (0.9% sodium chloride iv injection). Methylnaltrexone, at a dose of 0.3 mg/Kg, was administered diluted with 5 ml of normal saline as a single i.v. bolus over 1 minute followed by morphine (5-mg intravenous bolus). Then patients received iv morphine and a loading dose of ticagrelor. In this arm patients received placebo at visit 1. After a 7 ± 2 days wash-out period, patients crossed-over to the alternate study-treatment arm (methylnaltrexone).
  Placebo: Placebo will be administered as a 0.9% sodium chloride iv injection
  Morphine: After methylnaltrexone, patients will receive 5-mg intravenous morphine
  Ticagrelor: After morphine administration, patients will receive a 180-mg ticagrelor loading dose
Period: Visit 1
Arm/Group | Methylnaltrexone First | Placebo First
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Visit 2
Arm/Group | Methylnaltrexone First | Placebo First
Started | 14 (One subject completed visit 1 and then withdrew from the study for an adverse event (nausea).) | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Whole Study Population: Patients were randomly assigned in a 1:1 fashion to receive either i.v methylnaltrexone or placebo (0.9% sodium chloride iv injection). Methylnaltrexone, at a dose of 0.3 mg/Kg, was administered diluted with 5 ml of normal saline as a single i.v. bolus over 1 minute followed by morphine (5-mg intravenous bolus). Then patients received iv morphine and a loading dose of ticagrelor. After a 7 ± 2 days wash-out period, patients crossed-over to the alternate study-treatment arm.
Arm/Group | Whole Study Population
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Measured by VerifyNow P2Y12
Description: Platelet reactivity measured by VerifyNow P2Y12 2 hours after ticagrelor loading dose and reported as P2Y12 reaction units (PRU)
Time Frame: 2 hours
Measure: Least Squares Mean (95% Confidence Interval); unit: PRU
Groups:
- Methylnaltrexone; Placebo: Patients were randomly assigned in a 1:1 fashion to receive either i.v methylnaltrexone or placebo (0.9% sodium chloride iv injection). Methylnaltrexone, at a dose of 0.3 mg/Kg, was administered diluted with 5 ml of normal saline as a single i.v. bolus over 1 minute followed by morphine (5-mg intravenous bolus). Then patients received iv morphine and a loading dose of ticagrelor. After a 7±2 days wash-out patients received the alternate treatment.
  Treatment effects were evaluated comparing the functional parameters observed in the overall patient population after methylnaltrexone therapy with those achieved after placebo therapy regardless of the sequence in which patients received treatment.
Arm/Group | Methylnaltrexone | Placebo
Number analyzed (Participants) | 30 | 29
PRU | 130 [84 to 176] | 97 [59 to 136]
Statistical Analysis 1: Comparison: Methylnaltrexone vs Placebo; Test type: Superiority; p = 0.261, Mixed Models Analysis; Mean Difference (Final Values) = -32, 95% CI 2-sided [-90 to 25]

2. Secondary Outcome: Platelet Reactivity Measured by VASP
Description: Platelet reactivity measured by VASP 2 hours after ticagrelor loading dose and reported as platelet reactivity index (PRI)
Time Frame: 2 hours
Measure: Least Squares Mean (95% Confidence Interval); unit: PRI
Arm/Group | Methylnaltrexone | Placebo
Number analyzed (Participants) | 30 | 29
PRI | 47 [33 to 60] | 40 [29 to 51]

3. Secondary Outcome: AUC of Ticagrelor Plasma Levels
Description: The area under the plasma concentration vs. time curve from time 0 to the last measurable concentration (AUC) was calculated based on ticagrelor plasma levels
Time Frame: 6 hours
Measure: Geometric Mean (Full Range); unit: ng*hr/mL
Arm/Group | Methylnaltrexone | Placebo
Number analyzed (Participants) | 30 | 29
ng*hr/mL | 2952 [250 to 10133] | 2276 [24 to 7986]

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Methylnaltrexone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 8/30 | 10/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylnaltrexone (N=30) | Placebo (N=29)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)
nausea/vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
hypotension (Cardiac disorders) | 1 (1) | 0 (0)
dizziness (Cardiac disorders) | 0 (0) | 1 (1)
hypertensive urgency (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes